CLINICAL TRIAL: NCT03600103
Title: Technology Based Community Health Nursing to Improve cART Adherence and Virologic Suppression in Youth Living With HIV (TECH-N 2 CHECK-IN): A Regional Multi-site Study
Brief Title: Technology Based Community Health Nursing to Improve Combination Anti-Retroviral Therapy (cART) Adherence and Virologic Suppression in Youth Living With HIV
Acronym: Tech2Check
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00161462; 1R01MD011770-01 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-07-26 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections; Adherence, Medication
Keywords: adolescent; community health nursing; text messaging; mobile health
MeSH Terms: conditions — HIV Infections; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive standard of care.
- Intervention (Experimental): TECH2CHECK involves field visits by a CHN trained in disease intervention protocols, including clinical assessment, case management, counseling, and a behavioral intervention coupled with text messaging support for medication and self-care reminders.
  Interventions: Behavioral: Tech2Check

INTERVENTIONS:
Behavioral: Tech2Check — The intervention uses behaviors to improve HIV adherence and self-care. Investigators will use the Center for Disease Control (CDC) Partnership for Health (PfH) Medication Adherence.The CHN will administer PfH at all home/venue-based encounters, using communication styles that are more receptive to adolescents and young adults. Resources will be provided. At the end of the session, the participant will be able to state/demonstrate: goals of HIV care and adherence, meaning of CD4 and Viral Load (VL) measurements and the significance of their own measurements,signs of complications or problems for which participants need to seek additional care,understanding of optimal self-care.Further, CHNs will also provide tips to stay on schedule with taking their ART and problem-solve adherence barriers.
  Arms: Intervention

SUMMARY:
Human immunodeficiency virus (HIV) infection has disproportionately persisted as a public health threat to adolescents and young adults (AYA) from minority communities in the United States. HIV has evolved into a chronic disease, which can be managed in the outpatient setting with antiretroviral therapy (ART) designed to achieve virologic suppression and life expectancy equivalent for uninfected individuals. Community health nurse (CHN) interventions have been shown to increase access to appropriate resources, enhance health care utilization, and promote risk-reducing behavior among AYA. Use of short messaging service (SMS) messaging can further enhance clinical care by improving attendance at medical visits, medication adherence, and communication with the health care team.Investigators have used these two modalities in randomized trials of youth with complex sexually transmitted infections (STIs) in low-income minority communities with high feasibility and acceptability amongst AYA and families, remarkable improvements in visit completion, medication adherence, and reduction in recurrent STIs. The overarching goal of this project is to build on the evidence from this trial and to re-purpose the intervention for Young people living with HIV (YLHIV) in the same community who are having challenges with care and medication non-adherence.Investigators aim to compare the effectiveness of a technology-enhanced community health nursing intervention (TECH2CHECK) to a standard of care control group using a randomized trial design. The central hypothesis is that the intervention will result in higher rates of adherence to ART and virologic suppression. Investigators have demonstrated investigators' interdisciplinary team's capacity to follow urban AYA in the community, utilizing the combination of CHNs and outreach workers to optimize care according to national standards. TECH2CHECK aims to enroll 120 YLHIV followed at clinics specializing in HIV care in the Baltimore-Washington Metropolitan area and Jacksonville, Florida who are challenged with treatment adherence and randomizing participants to receive TECH2CHECK vs. standard of care. Results of this trial will inform best practices for engaging YLHIV by addressing the distal component of the continuum, critical to achieving the elusive 90-90-90 HIV goals.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants should be aged 12-25 years old diagnosed with HIV
* Eligible for ART, VL>20 copies/ml
* English speaking (>95% current clinic population)
* Aware of their HIV status
* Permanently reside in the Baltimore/Washington Metropolitan area or Jacksonville, Florida
* Willing to sign informed consent (including allowing communication with the participant's primary care provider). Informed consent includes being willing to complete study procedures; including randomization and community-based follow-up by our team.

Exclusion Criteria:

* Mental health, cognitive, or behavioral dysfunction that in the opinion of the site PI would impair effective participation
* Severe illness requiring hospitalization at the time of enrollment. This will be assessed at the team meetings designed to generate referrals.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Viral suppression | 18 months
  Viral suppression will be assessed by measuring plasma HIV-1 RNA (copies/mL). Viral suppression is defined as a viral load <20 copies/mL.

SECONDARY OUTCOMES:
Management Cost difference | 18 months
  To compare the cost of TECH2CHECK as compared to Standard of Care (SOC) for management of HIV in the outpatient setting. The costs of administering the different components of TECH2CHECK intervention and the standard of care will be based on a combination of direct observations, project records, and clinic invoices. The amount of staff and patient time (e.g. hours worked for CHN, patient transportation/visit time), consumable supplies (including miles traveled, antiretroviral costs, SMS costs, etc.), and equipment utilized (e.g., cell phones) for the intervention and SOC will be collected. Costs related to other health service utilization will be derived from ACASI, care utilization data.
Adherence to care as assessed by patient visits | 18 months
  We will examine attendance to clinical visits (proportion of appointments attended/appointments scheduled). This will be based on a binary (Yes/No) response to a questionnaire given out to patients.
Adherence to care as assessed by HRSA retention measure | 18 months
  We will also assess whether patients meet the Health Resources and Services Administration (HRSA) retention measure (2 provider visits in a 12-month period, with one appointment in each 6 month period, separated by at least 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Agwu, MD,ScM, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Florida, Jacksonville, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agwu AL, Yusuf HE, D'Angelo L, Rathore M, Marchesi J, Rowell J, Smith R, Toppins J, Trexler C, Carr R, Johnson B, Selden AK, Mahmoudi S, Black S, Guadamuz J, Huettner S, Trent M. Recruitment of Youth Living With HIV to Optimize Adherence and Virologic Suppression: Testing the Design of Technology-Based Community Health Nursing to Improve Antiretroviral Therapy (ART) Clinical Trials. JMIR Res Protoc. 2020 Dec 11;9(12):e23480. doi: 10.2196/23480. PMID 33306036